CLINICAL TRIAL: NCT06322589
Title: Evaluation of Human Efficacy of SOD Like Super Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMUH112-REC3-175
Record Dates: First submitted 2024-02-29; First posted 2024-03-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Dermatology
Keywords: Skin analysis; Skin care products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: placebo drink
- SOD like Super Drink (Experimental)
  Interventions: Dietary Supplement: SOD like Super Drink

INTERVENTIONS:
Dietary Supplement: SOD like Super Drink — consume 1 bottle per day
  Other Names: AVON SOD like Super Drink
  Arms: SOD like Super Drink
Dietary Supplement: placebo drink — consume 1 bottle per day
  Arms: placebo drink

SUMMARY:
To assess the efficacy of SOD like Super Drink on anti-oxidant capacity, immuno regulation and skin for human

ELIGIBILITY:
Inclusion Criteria:

* healthy adults aged between 30-65 years old

Exclusion Criteria:

* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder
* Patients with diseases of the skin, liver, kidney.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure (> 3 hr/week) in the past 4 weeks.
* Students who are currently taking courses taught by the principal investigator of this trial.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
the volume of skin wrinkles | Volume change from Baseline skin wrinkles at 8 weeks
  IRV full-face skin analyzer was utilized to measure skin wrinkles. Units: arbitrary units
the roughness of skin texture | Rating skin roughness from Baseline skin texture at 8 weeks
  IRV full-face skin analyzer was utilized to measure skin texture. Units: arbitrary units
the change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  Cutometer® was utilized to measure skin elasticity. Units: arbitrary units
the change of Total Anti-oxidative Capacity (TAC) of blood | Change from Baseline TAC at 8 weeks
  venous blood was sampled to measure TAC
the change of Superoxide Dismutase (SOD) of blood | Change from Baseline SOD at 8 weeks
  venous blood was sampled to measure SOD
the change of Glutathione S-transferase (GST) of blood | Change from Baseline GST at 8 weeks
  venous blood was sampled to measure GST
the change of Glutathione (GSH) of blood | Change from Baseline GSH at 8 weeks
  venous blood was sampled to measure GSH
the change of Malondialdehyde (MDA) of blood | Change from Baseline MDA at 8 weeks
  venous blood was sampled to measure MDA
the change of immune-related cytokines of blood | Change from Baseline immune-related cytokines at 8 weeks
  venous blood was sampled to measure immune-related cytokines

SECONDARY OUTCOMES:
the change of skin surface hydration | Change from Baseline skin surface hydration at 8 week
  Corneometer® CM 825 was utilized to measure skin surface hydration. Units: arbitrary units
the change of skin Transepidermal Water Loss (TEWL) | Change from Baseline TEWL at 8 week
  Tewameter® TM 300 was utilized to measure TEWL. Units: arbitrary units
the change of Skin Melanin Index | Change from Baseline skin Melanin Index at 8 week
  Mexameter® MX 18was utilized to measure Melanin Index. Units: arbitrary units
the change of Skin Erythema Index | Change from Baseline skin Erythema Index at 8 week
  Mexameter® MX 18was utilized to measure skin Erythema Index. Units: arbitrary units

OTHER OUTCOMES:
The change of liver function biomarkers (AST, ALT) of blood | Change from Baseline liver function biomarkers at 8 weeks
  Venous blood was sampled to measure liver function biomarkers
The change of renal function biomarkers (creatinine, BUN) of blood | Change from Baseline renal function biomarkers at 8 weeks
  Venous blood was sampled to measure renal function biomarkers
The change of self-assessment skin condition and immuno condition | Change from Baseline skin condition and immunol condition at 8 weeks
  A self-assessment questionnaire was collected to evaluate skin condition and immunol condition，As for the evalutation of skin condition ,the higher score the better；As for evaluation of immunol condition , the higher score the worse

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Mei Chiang, Principal Investigator — China Medical University of department of cosmeceutics
Locations (1):
- China Medical University of department of cosmeceutics, Taichung, Taiwan